CLINICAL TRIAL: NCT05739500
Title: The Clinical Trial 01 to Evaluate the Effectiveness of MRI-based Computer Aided Diagnosis Software (V1) for Glioma Segmentation, Gene Prediction and Tumor Grading
Brief Title: MRI-based Computer Aided Diagnosis Software (V1) for Glioma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mingge LLC (Industry)
Collaborators: Huashan Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Zhifeng Shi, Prof., Huashan Hospital
Other Study IDs: MINGGE-SW-00001-V1-01
Record Dates: First submitted 2022-12-28; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Glioma; Primary Brain Tumor
MeSH Terms: conditions — Glioma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — no intervention, just observation

SUMMARY:
The goal of this multi-center clinical trial is to evaluate the effectiveness of MRI-based computer-aided diagnosis software (V1) for glioma segmentation, gene prediction, and tumor grading. Machine learning methods such as high-precision tumor segmentation and classification and discrimination modeling can further optimize the non-invasive molecular diagnosis and prognosis prediction. The main question it aims to answer is whether the software can predict the molecular type and the prognosis quickly and correctly. The results will be compared with the real-world clinical data double-blindly. Finally, form a set of user-friendly automatic glioma diagnosis and treatment systems for clinics.

DETAILED DESCRIPTION:
BACKGROUND:

The molecular type is crucial for surgical planning and post-operative treatment of glioma. MRI-based radiomics is an emerging technique that extracts unrevealed information including pathology, biomarkers, and genomics by using automated high-throughput extraction of a large number of quantitative features. With the help of artificial intelligence, MRI-based radiomics could be a promising noninvasive method to reveal molecular type by using a quantitative radiomics approach for glioma.

AIM:

MRI-based computer-aided diagnosis software (V1) is an MRI-based radiomics tool with machine learning methods such as high-precision tumor segmentation and classification and discrimination modeling that can further optimize the non-invasive molecular diagnosis and prognosis prediction. The main question it aims to answer is whether the software can predict the molecular type and the prognosis quickly and correctly.

PROCESS:

Participants will read an informed consent agreement before surgery and voluntarily decide whether or not to join the experimental group. They will undergo preoperative multimodal magnetic resonance imaging, which is the routine neuro-images of preoperative evaluation. After surgery, the patient's tumor tissue samples will undergo specialist genetic testing to obtain multiple molecular diagnostic results, such as isocitrate dehydrogenase (IDH), telomerase reverse transcriptase promoter (TERTp), the short arm chromosome 1 and the long arm of chromosome 19 (1p/19q), et al. The participants need to be followed up for 1-year after surgery. Also, their imaging data, genotype data, clinical history data, pathology data, and clinical follow-up data will be analyzed for the study.

The preoperative Multimodality imaging will be input to the software (V1), and glioma segmentation, gene prediction, tumor grading, and lifetime will be analyzed by the software. The results will be compared with the real-world clinical data double-blindly. In order to evaluate the estimation performance of the software, several indexes will be calculated including accuracy (ACC), sensitivity (SENS), and specificity (SPEC). Finally, form a promising set of user-friendly automatic glioma diagnosis and treatment systems for clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Age front 18 to 70 years old (not including threshold), gender is not limited;
2. Preliminary diagnosis of glioma patients and patients who plan to undergo surgical treatment;
3. Preoperative cranial MRI (T1, T2, T2 Flair, T1 enhanced GE company magnetic resonance package), tumor pathological examination (H&E section, Kuoran Gene Company package), acceptable follow-up and brain MRI scan;
4. The patient himself voluntarily participated and signed the informed consent in writing.

Exclusion Criteria:

1. Patients who only underwent biopsy rather than surgical tumor resection;
2. Postoperative pathologically confirmed non-glioma patients;
3. Patients with multiple glioma metastases or multiple gliomas;
4. Patients who died of complications in the early postoperative period;
5. The researcher believes that this researcher should not be included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Preliminary diagnosis of glioma patients and patients who plan to undergo surgical treatment
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11-23 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy rate | end of the study (one year after the surgery of the last participants).
  describing the number of correct cases predicted by the software as a proportion of the total participants. The accuracy rate has a value between 0 and 1, with higher values indicating a more reliable tool.

CONTACTS AND LOCATIONS:
Overall Officials: Zhifeng Shi, MD., Principal Investigator — Huashan Hospital
Locations (1):
- Zhen Fan, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia CR, Slone SA, Dolecek TA, Huang B, Neltner JH, Villano JL. Primary central nervous system tumor treatment and survival in the United States, 2004-2015. J Neurooncol. 2019 Aug;144(1):179-191. doi: 10.1007/s11060-019-03218-8. Epub 2019 Jun 28. PMID 31254264
- [Background] Reardon DA, Wen PY. Glioma in 2014: unravelling tumour heterogeneity-implications for therapy. Nat Rev Clin Oncol. 2015 Feb;12(2):69-70. doi: 10.1038/nrclinonc.2014.223. Epub 2015 Jan 6. PMID 25560529
- [Background] Gillies RJ, Kinahan PE, Hricak H. Radiomics: Images Are More than Pictures, They Are Data. Radiology. 2016 Feb;278(2):563-77. doi: 10.1148/radiol.2015151169. Epub 2015 Nov 18. PMID 26579733
- [Background] Yu J, Shi Z, Lian Y, Li Z, Liu T, Gao Y, Wang Y, Chen L, Mao Y. Noninvasive IDH1 mutation estimation based on a quantitative radiomics approach for grade II glioma. Eur Radiol. 2017 Aug;27(8):3509-3522. doi: 10.1007/s00330-016-4653-3. Epub 2016 Dec 21. PMID 28004160